CLINICAL TRIAL: NCT05513469
Title: Biomarker Identification of Radionuclide Therapy-induced Radiation Responses
Acronym: Radio-Marker
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, M.N. Becx, PhD-student / coordinating investigator, Erasmus Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 80190
Record Dates: First submitted 2022-08-11; First posted 2022-08-24 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Neuroendocrine Tumors
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — lutetium Lu 177 dotatate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Peptide receptor radionuclide therapy (Other): PRRT 4x7.4GBq
  Interventions: Drug: Lutathera

INTERVENTIONS:
Drug: Lutathera — regulair PRRT of 4 cycles with 7.4GBq
  Other Names: 177lu-dotatate

SUMMARY:
Peptide receptor radionuclide therapy (PRRT) with [177Lu]Lu-DOTA-[Tyr3]octreotate (177Lu-DOTATATE) is a form of internal radiation treatment for patients with neuroendocrine tumors (NET) to reduce tumor growth and stabilize disease. Due to limited response rates, there is a need to improve this therapy. A better understanding of therapeutic radiobiological responses, such as transcriptional and DNA damage responses, could contribute to identification of biomarkers for toxicity and/or efficacy prediction. Easy access to biological samples for biomarker discovery would be via a so-called liquid biopsy (drawing blood) to collect healthy peripheral blood mononuclear cells (PBMCs) or circulating tumor DNA (ctDNA) for further investigation.

Exposure to ionizing radiation (IR) such as by PRRT leads to complex cellular responses including activation of the DNA damage response and changes in gene expression which can differ between individuals. This was previously shown for ex vivo external beam radiation of blood cells in which radiation responsive genes were identified. These genes were also similarly up- or downregulated following in vivo exposure to total-body irradiation of patients. In addition, different studies have shown a good correlation between radiation dose to the blood and DNA double strand break induction in PBMCs for various PRRT-like treatments. These results show that such events can be measured in PBMCs and indicate that ex vivo irradiation can mimic the in vivo transcriptional regulation and DNA damage induction. Therefore, to identify PRRT-induced cellular responses, the investigators will analyze the effects of 177Lu-DOTATATE IR on the transcriptional regulation in PBMCs and compare this regulation to radiation dose and DNA damage induction.

In addition, it was shown that levels of ctDNA can be associated with treatment response and anticancer treatment is also shown to influence ctDNA methylation patterns. The investigators will therefore explore dynamics of ctDNA levels and methylation patterns before and after PRRT to provide more knowledge of the effect of radiation response on ctDNA.

This is a pilot study to validate the possibility of determining the radiation response of PRRT with 177Lu-DOTATATE in PBMCs and ctDNA.

DETAILED DESCRIPTION:
Altogether, the PBMC and ctDNA analyses will provide essential information on the PRRT radiation response using blood as easily accessible material. Future research can focus on development of radiation response biomarkers based on the outcomes of this study.

Objective: This is a pilot study to validate the possibility of determining the radiation response of PRRT with 177Lu-DOTATATE in PBMCs and ctDNA.

Study design: Prospective translational study with additional blood collections at 4 timepoints during regular patient care for ex vivo characterisation.

Study population: Twenty patients with locally advanced or metastatic NET receiving the first PRRT cycle of 7.4 GBq 177Lu-DOTATATE.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

Participants who receive standard PRRT will undergo 4 additional venipunctures during their scheduled stay in the hospital for PRRT administration. The burden of the venipunctures is minimal. There is no benefit for particitants.

ELIGIBILITY:
Inclusion Criteria:

* Patient with an advanced, well-differentiated midgut neuroendocrine tumor.
* Indication for treatment with PRRT with 7.4 GBq 177Lu-DOTATATE as determined by the multidisciplinary team.
* Age ≥ 18 years.

Exclusion Criteria:

* Failure to obtain informed consent.
* Patient received IR for imaging purposes within one week prior to PRRT or IR for therapeutic purposes within 3 months prior to PRRT.
* Previous treatment with PRRT.
* Indication to receive another activity of PRRT than 7.4 GBq.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Transcriptional regulation and DNA damage induction in PBMCs after PRRT. | 2 years
  DNA damage will be assessed by immunofluorescent stainings and microscopic detection of γ-H2AX and 53BP1 RIF. RIF numbers of at least 50 cells from at least 4 fields of view per blood sample will be quantified using an automated quantification macro in ImageJ.
  RNA isolation, sequencing, analysis and qPCR validation will be done. Validation of the identified differentially expressed genes will be performed in triplicate by qPCR. For sequencing, we will use an unique in-house analysis method using a Snakemake pipeline. RIF and sequencing analysis will be performed on blinded samples to perform unbiased analysis.

SECONDARY OUTCOMES:
mimic transcriptional regulation and DNA damage induction in PRRT ex vivo. | 2 years
  Untreated blood from the patient will be treated with 177Lu-DOTATATE ex vivo. Analysis of transcriptional regulation and DNA damage induction will be done as mentioned in the description of outcome 1.
detection of ctDNA in NET patients | 2 years
  For the assessment of circulating biomarkers of the tumor cells we will measure ctDNA levels in the blood.

OTHER OUTCOMES:
Evaluate the effect of PRRT on ctDNA levels. | 2 years
  ctDNA levels will be measured in the blood before PRRT and 8 weeks after the first cycle.
methylation sequencing ctDNA | 2 years
  DNA methylation sequencing method will be used to analyze the ctDNA. The MeD-seq assay will be used for genome-wide DNA methylation profiling on cell-free DNA (cfDNA)

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus MC, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No